CLINICAL TRIAL: NCT02639039
Title: Cortisone Injection vs Trigger Point Dry Needling Fin the Treatment of Greater Trochanter Pain Syndrome: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110495
Record Dates: First submitted 2015-12-02; First posted 2015-12-24 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries | interventions — Cortisone; Steroids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cortisone Injection (Active Comparator): Fifty patients with GTPS will be randomized into a CI or TDN group. Treatment will be carried out at the 1st visit following consent according to SOC. Treatment will be administered according to standard of care for up to 6 weeks.
  Interventions: Drug: Cortisone Injection
- Trigger Point Dry Needling (Active Comparator): Fifty patients with GTPS will be randomized into a CI or TDN group. Treatment will be carried out at the 1st visit following consent according to SOC. Treatment will be administered according to standard of care for up to 6 weeks.
  Interventions: Procedure: Trigger Point Dry Needling

INTERVENTIONS:
Drug: Cortisone Injection — Exact location and technique of injection within the region of the involved greater trochanter will be determined by the provider. The number of f/u visits within 6 wks following initiation of treatment will be determined by the provider, but CI is the only treatment.
  Other Names: Steroid injection
  Arms: Cortisone Injection
Procedure: Trigger Point Dry Needling — Exact location of needle insertion, technique and number of penetrations within the region of the involved posterolateral hip will be determined by the provider. The number of f/u visits within 6 wks following initiation of treatment will be determined by the provider, but TDN is the only treatment.
  Arms: Trigger Point Dry Needling

SUMMARY:
The purpose of this study is to determine if trigger point dry needling (TDN) is as effective as cortisone injection (CI) in reducing pain and improving function in patients with greater trochanteric pain syndrome (GTPS).

DETAILED DESCRIPTION:
This study aims to investigate the potential of TDN as an effective alternative to CI for patients with GTPS by directly comparing pain and functional outcomes of patients receiving TDN or CI for the treatment of GTPS over a 6 week period. The investigators hypothesize that patients treated with TDN will be equally improved in pain and function as those treated with CI. If TDN is demonstrated to be equally or more effective than steroid injection in this pilot study, then the investigators have the basis to launch larger studies. Ultimately, the investigators want to determine if TDN is an effective treatment alternative for GTPS for providers and patients who want to avoid the potential detrimental side-effects of steroids.

Approach: Prospective, randomized, partially-blinded design

Aim: To determine if administration of TDN is as effective as CI in reducing lateral hip pain and improving function in patients diagnosed with greater trochanteric pain syndrome. The investigators expect to demonstrate effectiveness of TDN in the treatment of GTPS to a degree that is equal to CI. Doing so would prompt further outcomes research for TDN. Supportive research and subsequent clinical acceptance of TDN as a primary treatment for this condition would offer an alternative to patients who want or need to avoid steroids.

Based on the literature, this is the first study to investigate the effectiveness of TDN in the treatment of GTPS and directly compare pain and functional outcomes of patients receiving TDN versus CI for the treatment of GTPS.

Methods. Fifty patients with GTPS will be randomized into a CI or TDN group. Treatment will be administered according to standard of care for up to 6 weeks. Numerical pain and functional ratings for each patient will be collected at 0, 1, 3, and 6 weeks of treatment. Data analysis will determine if TDN is as effective as cortisone.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* lateral hip pain (anywhere from iliac crest to mid ITB)
* active email account

Exclusion Criteria:

* low back pain associated with the hip pain
* motor and/or sensory impairment consistent with radiculopathy
* active infection/malignancy of the hip
* connective tissue disease
* pregnancy
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Participants change in pain rating scores from baseline to 6 weeks will be accessed. | Baseline and 6 weeks
Patient specific function score (PSPS) from baseline to 6 weeks will be accessed. | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kindyle L Brennan, PhD, Principal Investigator — Orthopedic Therapist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brennan KL, Allen BC, Maldonado YM. Dry Needling Versus Cortisone Injection in the Treatment of Greater Trochanteric Pain Syndrome: A Noninferiority Randomized Clinical Trial. J Orthop Sports Phys Ther. 2017 Apr;47(4):232-239. doi: 10.2519/jospt.2017.6994. Epub 2017 Mar 3. PMID 28257614